CLINICAL TRIAL: NCT02217397
Title: Combinations of Oral Appliance and CPAP for Patients With Severe Obstructive Sleep Apnea Untolerate High-pressure CPAP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Principal Investigator, National Taiwan University Hospital, Seep cencer, National Taiwan University Hospital, National Taiwan University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201402033RINC
Record Dates: First submitted 2014-08-05; First posted 2014-08-15 (Estimated); Last update posted 2015-03-18 (Estimated); Status verified 2014-08

CONDITIONS: Obstructive Sleep Apnea
Keywords: Apnea-hyponea Index, CPAP, Obstructive Sleep Apnea, Oral Appliance
MeSH Terms: conditions — Sleep Apnea, Obstructive; Microcephaly, Primary Autosomal Recessive, 6 | interventions — Continuous Positive Airway Pressure; Combined Modality Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- OA, CPAPm, combination therapy (Experimental)
  Interventions: Device: OA, CPAP, combination therapy

INTERVENTIONS:
Device: OA, CPAP, combination therapy

SUMMARY:
Obstructive sleep apnea (OSA) is a situation of repetitive upper airway obstruction during sleep. For patients with severe OSA, continuous positive airway pressure (CPAP) therapy was the standard therapy, especially those with daytime sleepiness and cardiovascular comorbidities. Although CPAP is effective in OSA treatment, the poor adherence due to high pressure was often reported. Instead, oral appliance (OA) was the alternative for those who could not tolerance CPAP or mild to moderate OSA. Oral appliance was less effective in compared with CPAP, but OA is more tolerable and acceptable in OSA patients.

Only one observation study addressed the effects of the combinations of OA and CPAP in OSA patients . The pilot study displayed combination therapy of CPAP and OA is effective in OSA patients and could decrease CPAP pressure. However, the study enrolled the patients with CPAP intolerance according to the subjective chief complaint, not the objective CPAP pressure data. In the present study, we studied the effects of combinations of CPAP and OA for patients with severe OSA who could not tolerate CPAP with high-pressure setting.

DETAILED DESCRIPTION:
This is a prospective study in a tertiary teaching hospital, National Taiwan University Hospital. Patients are eligible with age ≧ 20 years old, severe OSA [apnea-hyponea index (AHI) >= 30/hr] who could not tolerate CPAP pressure >15 cmH2O, determined by manual titration (first titration) and willing to use OA.

The study designed was found out the patients with severe OSA (AHI >= 30/hr ). With first titration, the investigators excluded the severe OSA patients using CPAP (CPAP pressure < 15 cmH2O) and could tolerate CPAP. Those patients who could not tolerance CPAP high pressure setting started a three-month oral appliance trial. Then, the investigators repeated the full-channel polysomnography (PSG) with second titration on those with residual AHI ≧ 10/hr while patients were on OA. Therefore, those patients treated with combinations of OA and CPAP for three months and then repeated the PSG. The washout period in each therapy was two weeks. The total follow-up period is about 6 months after enrolled.

The investigators collected the demographic data from medical records and PSG data, including age, gender, body mass index (BMI), CPAP titration, AHI, total sleep time, oxygen desaturation, and arousal index…et al.

Our primary end point is the changes in AHI compared with combination therapy, and OA use. The secondary end points are the difference in titrated CPAP pressure, BMI, blood pressure, and daytime sleepiness compared with combination therapy and OA use.

Statistics analysis Data are presented as mean ± standard deviation (SD). Continuous variables were tested by paired Student's t test in group comparisons. Statistical significance was assumed when a null hypothesis could be rejected at p<0.05. The investigators compared the difference between combination therapy, OA, and baseline by ANOVA, repeated measure. Statistical analysis was done using the SPSS 22.0 for Windows.

ELIGIBILITY:
Inclusion Criteria:

1. New diagnosed obstructive sleep apnea patients older than 20 years old
2. AHI more than 30/hr with moderate to severe obstructive sleep apnea
3. Willing to accept CPAP and OA treatment

Exclusion Criteria:

1. nasal problems causing CPAP intolerance
2. status post uvulopalatopharyngoplasty
3. alcohol abuse and dependence
4. life expectancy less than 6 months
5. severe cardiopulmonary distress.

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2014-08; Primary Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
The difference of AHI (Apnea Hypopnea Index ) in different treatment (baseline, OA, combination therapy) | baseline and1, 3, 6 months later
  The participants will be followed every month over out patient clinic with measures of change with AHI, sleep quality of life with different treatment (baseline, OA, combination treatment group).
  The investigators will record the AHI in different treatment group with OA, CPAP or combination therapy and read if AHI decreased after combination therapy use.

CONTACTS AND LOCATIONS:
Overall Officials: Peilin Lee, PhD, Study Director — Center of Sleep Disorder, National Taiwan University Hospital